## CONSENT FORM FOR TEACHER PARTICIPATION IN HUMAN RESEARCH AT MONTANA STATE UNIVERSITY

**PROJECT TITLE**: A Trauma-Informed Intervention for Positive Youth Development and Teacher Wellness in Rural Montana

INVESTIGATOR: Lauren Davis, Assistant Professor, Montana State University

RATIONALE FOR THE RESEARCH: We would like to invite you to participate in a research project to learn about how certain activities might help relieve your stress and improve your quality of life and job satisfaction. We are asking for your help because we don't know very much about how to best support teacher wellbeing, which in turn supports student wellbeing and achievement. Participation in this study is completely voluntary. If you agree to participate in our study, we are going to ask you to answer some questions about your stress levels, career satisfaction, and overall wellbeing before and after this 6-week program. We want to know if certain activities help reduce your stress—specifically, yoga. Here's what the program will look like:

\*Yoga: Each session will highlight deep breathing, mindful movement, and stress relief. Sessions will begin with goal-setting, will move into the physical practice, and will end with a peaceful reflection that will help you feel less stressed. This program will take place twice weekly, online and synchronously, for 6 weeks. You may have students participating in a student-version of this program at the same time as you during their physical education class and/or online.

At the end of the program, we may ask you if you feel like you are less burned out at work, if you feel less stressed out, or if you feel happier or less anxious. In order to measure your stress levels, your stress hormone (cortisol) levels will be tested throughout the program through a collected saliva (spit) sample; you can learn more about the procedure for this safe, non-invasive process here:

https://www.nationwidechildrens.org/family-resources-education/health-wellness-and-safety-resources/helping-hands/saliva-cortisol-test-collection-guidelines. We will also be measuring your resting heart rate variability with a sensor at three points during the study. As an incentive for your participation, if you complete all of the study activities, you will be eligible to receive payment for each class session in the form of a gift card, as well as a gift card for completing all surveys. Because of our budget, we are limiting participation to the first 40 teachers to sign up for the study. You can ask questions about the details of study at any time. If you decide at any time not to continue participating, then you won't be a part of the study.

The questions we will ask are only about what you think and feel before and after the study, which will take place for 6 weeks. There are no right or wrong answers; this is not a test. We will also ask you to write down and share with your reactions to the yoga sessions in an online journal each week so we can learn what was helpful to you in this study

**PROCEDURES:** Participation is voluntary. If you agree to participate, the confidential survey data you provide will be used in the study, and your responses will be kept anonymous. You will also be eligible for participation incentives (see below).

RISKS OF PARTICIPATION: It is possible that the program may bring up strong feelings for you; it's important for you to know your own limits and take care of yourself during the program. If you ask or if you need it, we will give you information for where you can find extra support. Some examples are:

- Talking with someone who you can trust
- Calling 911, your doctor or other healthcare provider

- Going to an Emergency Room Calling 1-800-273-TALK (8255) to talk with a crisis worker for free
- Texting 741741 to text with a counselor for free
- Visiting NowMattersNow.org to learn skills for dealing with thoughts of suicide

**BENEFITS OF PARTICIPATION:** Importantly, there are also potential benefits to being part of the study. You may have reductions in severity of depression and/or anxiety as well as improvements in overall behavioral health and well-being. Additional benefits for participants may be improved sleep, improved social skills, improved emotion regulation, and improvements in career satisfaction and/or burnout.

CONFIDENTIALITY: All research information will be kept confidential. All information will be kept in a secure platform that is accessible only to the researchers by password and institutional credentials. This information will be saved as long as it is scientifically useful; typically, such information is kept for five years after publication of the results. Results from this study may be presented at professional meetings and in publications. You will not be identified individually.

| COMPENSATION: Teacher incentives for participation in the study will be in the form of a gift card at the rate of \$15 per yoga class (limit of 12 classes total). Additional gift cards of \$50 will be offered for completion of pre- and post-surveys during the study. |
|---|
| I,, have read and fully understand this consent form. I sign it freely and voluntarily. I hereby give permission for my participation in this study and understand that I may withdraw from the study at a later time. I have received a copy of this consent form. Signature of Participant |
| Date |

Contact Information: Dr. Lauren Davis (Principal Investigator) Montana State University Lauren.davis6@montana.edu 406-994-7424

Note: This form is a requirement of Montana State University's Institutional Review Board (IRB). An IRB is an administrative body established to protect the rights and welfare of human research subjects recruited to participate in research activities conducted by faculty members of Montana State University. The IRB is charged with the responsibility of reviewing, prior to its initiation, all research involving human participants. The IRB is concerned with protecting the welfare, rights, and privacy of human subjects and has the authority to approve, disapprove, monitor, and require modifications in all research activities that fall within its jurisdiction as specified by both the federal regulations and institutional policy. If you have any questions regarding this proposed project, their contact information is listed below; please don't hesitate to reach out to them with any concerns. Montana State University Institutional Review Board Mark Quinn, Chair P.O. Box 173610 Bozeman, MT 59717

## **Student Assent Form (Experimental)**

We are doing a research project to learn about how certain types of activities might help lower your stress and make your life better. We are asking for your help because we don't know very much about how kids your age are best able to reduce their stress levels.

If you agree to join our project, we are going to ask you some questions about yourself and your stress levels before and after this 6-week program. We want to know if you feel like certain activities help you feel calmer and/or happier after participating in yoga. Here's what the activities might look like:

\*Yoga: Each session will highlight deep breathing, mindful movement, and stress relief. Sessions will begin with goal-setting, then the physical practice, and will end with a peaceful relaxation activity that will help you feel less stressed. This will take place twice weekly for 6 weeks during your physical education class and/or online.

After you complete the program, we may ask you if you feel more focused in class, if you feel less stressed out, or if your grades have changed with the exercise program. We will also be collecting a sample of your saliva (spit) periodically during the program to measure your stress hormone levels (cortisol) to see if this program helps reduce your stress. We will also be measuring your resting heart rate variability with a sensor at three points during the study. As an incentive for your participation, if you complete all of the study activities, you will get a free Fitbit health tracker at the end of the study!

The questions we will ask you are only what you think before and after the study. There are no right or wrong answers, and this is not a test--it will NOT have any impact on your school grades. As a part of the research project, we will look at some information on your student records, your stress levels, and ask you to respond to a survey where you will provide the number of difficult life experiences you have experienced. To protect your privacy, no information concerning the details of these experiences will be collected other than the number you have experienced. All your information will be kept completely confidential and private. However, if you start to have suicidal thoughts, think about hurting yourself or others during any part of the study, we will let school officials know for your own and others' safety. You can ask questions about this study at any time. If you decide at any time not to finish, then you don't have to be a part of the study; participation in this study is completely voluntary.

The questions on the surveys we will ask are only about what you think. There are no right or wrong answers because this is not a test. We will also ask you to write down and share with us your reactions to the yoga session in a journal each week so we can learn what was helpful to you in this study. It is possible that the program may bring up strong feelings for you; it's important for you to know your own limits and take care of yourself during the program. If you ask or if you need it, we will give you information for where you can find extra support. Some examples are:

- Talking with someone who you can trust
- Calling 911, your doctor or other healthcare provider
- Going to an Emergency Room
- Calling 1-800-273-TALK (8255) to talk with a crisis worker for free
- Texting 741741 to text with a counselor for free
- Visiting NowMattersNow.org to learn skills for dealing with thoughts of suicide

Importantly, there are also potential benefits to being part of the study. Participants may have reductions in severity of depression and/or anxiety as well as improvements in overall behavioral health and well-being. Additional benefits for participants may be improved sleep, improved social skills, improved emotion regulation, improved academic behaviors and outcomes.

If you sign this paper, it means that you have read this and that YOU DO NOT WISH to be in the study. If you want to be in this study, don't sign this paper. Being in the study is up to you, and no one will be upset if you don't sign this paper or if you change your mind later. It also won't affect your grades or school standing whatsoever.

| Your signature: | |
|--------------------------|-------------------|
| Your printed name: | |
| Contact Information: | |
| Dr. Lauren Davis (Princi | pal Investigator) |

Note: This form is a requirement of Montana State University's Institutional Review Board (IRB). An IRB is an administrative body established to protect the rights and welfare of human research subjects recruited to participate in research activities conducted by faculty members of Montana State University. The IRB is charged with the responsibility of reviewing, prior to its initiation, all research involving human participants. The IRB is concerned with protecting the welfare, rights, and privacy of human subjects and has the authority to approve, disapprove, monitor, and require modifications in all research activities that fall within its jurisdiction as specified by both the federal regulations and institutional policy. If you have any questions regarding this proposed project, their contact information is listed below; please don't hesitate to reach out to them with any concerns.

Montana State University Institutional Review Board Mark Quinn, Chair P.O. Box 173610 Bozeman, MT 59717 Ph (406) 994-4707

Montana State University Lauren.davis6@montana.edu

406-994-7424

## **Parent Consent Form (Experimental)**

Parents and Guardians,

We would like to invite your child to participate in a research project to learn about how certain activities might help them relieve stress and improve their quality of life. We are asking for your child's help because we don't know very much about how students your child's age might be able to best cope with and reduce stress. Participation in this study is completely voluntary. If you agree to your child being in our study, we are going to ask your child to answer a few questions about their stress levels and overall well-being before and after this 6-week program. We want to know if certain activities help reduce their stress—specifically, yoga. Here's what your child's activities might look like:

\*Yoga: Each session will highlight deep breathing, mindful movement, and stress relief. Sessions will begin with goal-setting, will move into the physical practice, and will end with a peaceful reflection that will help students feel less stressed. This program will take place twice weekly during your child's regularly scheduled physical education class and/or online.

At the end of the program, we may ask your child if they feel like they can concentrate in class more, if they feel less stressed out, or if they feel happier or less anxious. In order to measure stress levels, students' stress hormone (cortisol) levels will be tested throughout the program through a collected saliva (spit) sample; you can learn more about the procedure for this safe, non-invasive process: <a href="https://www.nationwidechildrens.org/family-resources-education/health-wellness-and-safety-resources/helping-hands/saliva-cortisol-test-collection-guidelines">https://www.nationwidechildrens.org/family-resources-education/health-wellness-and-safety-resources/helping-hands/saliva-cortisol-test-collection-guidelines</a>. We will also be measuring your child's resting heart rate variability with a sensor at three points during the study. As an incentive for your child's participation, if they complete all of the study activities, they will get a free Fitbit health tracker at the end of the study! You or your child can ask questions about the details of study at any time. If you or they decide at any time not to continue participating, then they won't be a part of the study.

The questions we will ask are only about what your child thinks and feels before and after the study, which will take place for 6 weeks. There are no right or wrong answers, and we will explain to them that this is not a test. We will also ask your child to write down and share with us his or her reactions to the yoga session in a journal each week so we can learn what was helpful to them in this study. As a part of the study, we will look at your child's academic records and stress levels measured in multiple ways; specifically, we will examine their MAPS scores, attendance/tardiness records, and behavioral referrals before and after the study. We will also ask your child to fill out surveys that gather information about their overall quality of life, and we will also give students a survey where they will be providing the number of difficult life experiences they have experienced. In order to protect your child's privacy, no information concerning the details of these experiences will be collected other than the number the child has experienced. All student information will be kept completely confidential and private--random ID numbers will be assigned by your child's teacher to each child in the study. However, in the event that a child shows any indication of suicidal thoughts, risk of self-harm, or harm to others during any part of the study, we will promptly notify school officials to discuss appropriate responses. Copies of all surveys and questionnaires will be provided to parents/guardians by request prior to the beginning of the program.

It is possible that the program may bring up strong emotions for the participants; to help with this this, the research team will caution students that this may happen, and we will and emphasize the importance of self-care and knowing one's own limits with the program. If needed, referrals for additional, outside treatment will be provided if necessary and/or requested. Additional resources include:

- Talking with someone who you can trust
- Calling 911, your doctor or other healthcare provider
- Going to an Emergency Room
- Calling 1-800-273-TALK (8255) to talk with a crisis worker for free
- Texting 741741 to text with a counselor for free

Visiting NowMattersNow.org to learn skills for dealing with thoughts of suicide

Importantly, there are also potential benefits to being part of the study. Participants may have reductions in severity of depression and/or anxiety as well as improvements in overall behavioral health and well-being. Additional benefits for participants may be improved sleep, improved social skills, improved emotion regulation, improved academic behaviors and outcomes.

If you do NOT want your child to participate in this study, please return this form to the school immediately upon receipt. Being in the study is up to you and your child. No one will be upset if you don't want your child to be in the study or if you or your child decide later not to participate. It will also not impact your child's grades or school standing in any way. If you WANT your child to participate in the study, NO ACTION is needed on your part.

Please sign below if you do NOT want your child to participate:

| Your child's name: | |
|---|---|
| Your signature: | |
| Your printed name: | Date: |
| Contact Information: | |
| On Layman Davis (Dringinal Investigator) M | Santona Stata University I over devise@montona edv. 10 |

Dr. Lauren Davis (Principal Investigator) Montana State University; Lauren.davis6@montana.edu; 406-994-7424

<u>Note:</u> This form is a requirement of Montana State University's Institutional Review Board (IRB). An IRB is an administrative body established to protect the rights and welfare of human research subjects recruited to participate in research activities conducted by faculty members of Montana State University. The IRB is charged with the responsibility of reviewing, prior to its initiation, all research involving human participants. The IRB is concerned with protecting the welfare, rights, and privacy of human subjects and has the authority to approve, disapprove, monitor, and require modifications in all research activities that fall within its jurisdiction as specified by both the federal regulations and institutional policy. If you have any questions regarding this proposed project, their contact information is listed below; please don't hesitate to reach out to them with any concerns.

Montana State University Institutional Review Board Mark Quinn, Chair P.O. Box 173610 Bozeman, MT 59717 Ph (406) 994-4707